CLINICAL TRIAL: NCT02932709
Title: Effect of Telephone Follow-up on Repeated Suicide Attempt in Patients Discharged From an Emergency Psychiatry Department: a Controlled Study
Brief Title: Effect of Telephone Follow-up on Repeated Suicide Attempt in Patients
Acronym: EXBRAYAT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Groupement Régional de Santé Publique (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1008071; 2010-A00804-35 (Other: ANSM)
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Suicide, Attempted
Keywords: Emergency; follow-up; nurse; phone; suicide attempts
MeSH Terms: conditions — Suicide, Attempted; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients admitted of Psychiatry: Only patients who had a suicide attempt admitted to the Department of Emergency Psychiatry.
  Interventions: Behavioral: suicide attempt

INTERVENTIONS:
Behavioral: suicide attempt — suicide attempt : We evaluated the effectiveness of telephone follow-up of patients who had referred to an emergency psychiatric unit for attempted suicide on any further attempt/s over the following year.

SUMMARY:
Attempted suicide is a major public health problem, and the efficacies of current postvention protocols vary. The investigators evaluated the effectiveness of telephone follow-up of patients referred to an emergency psychiatric unit for attempted suicide on any further attempt/s over the following year.

In a single-center, controlled study with intent to treat, they evaluated the efficacy of a protocol of telephone follow-up of patients at 8, 30, and 60 days after they had been treated for attempted suicide. For comparison, they evaluated as controls patients with similar social and demographic characteristics referred to their emergency psychiatric unit in the year prior to the study who did not receive telephone follow-up after their initial hospitalization. Data were analyzed using logistic regression.

DETAILED DESCRIPTION:
The importance of suicide and suicidal attempts recurrence is a major public health problem. Indeed, the suicide attempt is one of the most important predictors of suicide, as well as suicidal relapse is considered a suicide risk factor. It is therefore essential to establish the suicidal relapse prevention devices.

Moreover, the consensus conference on suicidal crisis (6) in particular stresses the importance of organizing continuity of care and foster a therapeutic alliance to avoid a break in continuity of care.

This study aims to evaluate the effectiveness of telephone Callback patients on suicide rate of recurrence at 6 months of suicidal gesture. A secondary objective is to assess and promote compliance.

Patients were included after a psychiatric interview following a suicide attempt in the North hospital's emergency unit no emergency hospitalization or indication in the interview before the release of the psychiatric emergency service. The interview provides an assessment of suicide risk and oral information about the protocol. A map showing the coordinates of the psychiatric emergency service and a reminder of the protocol is given. A consent form is signed. This protocol does not replace the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* Patient who have attempted suicide regardless of the medium
* Patient falling 4 psychiatric sectors covered by the CHU of Saint-Etienne
* Major and minor Patient (with parental permission)
* Patient for which there is no evidence of psychiatric hospitalization sector or clinic immediately after switching to the suicidal act

Exclusion Criteria:

* Homeless Patient
* Patients for whom Callback is not possible (no phone, incarceration ...)
* Patient who do not speak French
* Patient admitted sector or clinic following the psychiatric interview inclusion
* Patient Refusal
* Medical Reason
* Deleterious character of recontact by a doctor of the psychiatric emergency after passing the act

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the Department of Emergency Psychiatry of CHU Saint-Etienne for suicide attempt
Sampling Method: Non-Probability Sample
Enrollment: 876 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Comparison of suicidal recurrence rate | 6 months
  Number of relapses of suicide attempts per patient over a period of 6 months.

SECONDARY OUTCOMES:
Assess the impact of the device on the number of deaths by suicide | 6 months
  Number of deaths by suicide

OTHER OUTCOMES:
Assess the impact on adherence to treatments | 6 months
  The rate of adherence to treatments
Measuring the time between the TS and the first recurrence | 6 months
  Time of recurrence compared to the suicide attempt

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France